CLINICAL TRIAL: NCT07129044
Title: The Effect of the Flipped Classroom Model on Nursing Students' Pediatric Pain Management Knowledge and Learning Motivation: A Randomized Controlled Trial
Brief Title: The Effect of the Flipped Classroom Model on Pediatric Pain Management Knowledge and Learning Motivation of Nursing Students
Acronym: FLIPNURSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Belli (Other)
Responsible Party: Sponsor-Investigator, Mustafa Belli, Assistant Professor, Department of Pediatric Nursing, Faculty of Health Sciences, Burdur Mehmet Akif Ersoy University, Burdur Mehmet Akif Ersoy University
Organization: Burdur Mehmet Akif Ersoy University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ErsoyU-Belli-FC2022; 1070 (Other: Ege University Health Sciences Scientific Research and Publication Ethics Committee)
Record Dates: First submitted 2025-08-04; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Pain Management
Keywords: Pediatric pain management; Flipped classroom; Nursing students; Learning motivation; Randomized controlled trial
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to either the intervention group receiving flipped classroom-based pediatric pain management training or the control group receiving self-directed learning. The intervention lasted four weeks, and data were collected at three time points: pre-test (baseline), post-test (immediately after the intervention), and follow-up (three months later).
Masking Description: Not applicable. Participants and researchers were aware of group assignments due to the nature of the educational intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flipped Classroom Training on Pediatric Pain Management (Experimental): Participants in this group received pediatric pain management training through a flipped classroom model for 4 weeks. Training videos and readings were provided in advance and in-class sessions included interactive activities, discussions, and case-based learning.
  Interventions: Behavioral: Flipped Classroom Training on Pediatric Pain Management
- Self-Directed Learning on Pediatric Pain Management (Active Comparator): Participants in this group received the same pediatric pain management materials as the intervention group (lecture notes, readings, and video lectures) for self-study without any interactive activities or instructor-led sessions.
  Interventions: Behavioral: Self-Directed Learning on Pediatric Pain Management

INTERVENTIONS:
Behavioral: Flipped Classroom Training on Pediatric Pain Management — Participants in this group received pediatric pain management training designed to increase nursing students' knowledge and motivation. The training was delivered using a flipped classroom model over 4 weeks. Students were provided with pre-class educational materials, including video lectures, readings, and lecture notes. In-class sessions included interactive activities, discussions, case-based learning, and problem-solving exercises. Content was based on current pediatric pain management guidelines and adapted to nursing education standards.
  Arms: Flipped Classroom Training on Pediatric Pain Management
Behavioral: Self-Directed Learning on Pediatric Pain Management — Participants in this group received pediatric pain management training designed to increase nursing students' knowledge and motivation. Students were provided with the same pre-class educational materials as the intervention group, including video lectures, readings, and lecture notes, for self-study without any interactive activities or instructor-led sessions. Content was based on current pediatric pain management guidelines and adapted to nursing education standards.
  Arms: Self-Directed Learning on Pediatric Pain Management

SUMMARY:
The aim of this randomized controlled trial was to evaluate the effect of the flipped classroom model on pediatric pain management knowledge and learning motivation among nursing students. A total of 84 third-year nursing students from a public university in Turkey were randomly assigned to intervention (n=42) and control (n=42) groups. The intervention group received education using the flipped classroom model, while the control group followed a self-directed learning approach.

Data were collected at three time points: before the intervention (pre-test), one month after the intervention (post-test), and three months after the intervention (follow-up test). The Pediatric Pain Knowledge Test and the Motivation Scale Towards Learning were used to assess outcomes.

At baseline, there were no significant differences between the groups. Post-test and follow-up results showed that the intervention group demonstrated a statistically significant and sustained increase in both pediatric pain knowledge and learning motivation scores (p<0.001), while the control group showed no meaningful change.

These findings support the flipped classroom model as an effective and sustainable teaching strategy in nursing education, particularly for improving knowledge and motivation in pediatric pain management.

DETAILED DESCRIPTION:
This randomized controlled trial aimed to evaluate the effectiveness of the flipped classroom model in enhancing nursing students' pediatric pain management knowledge and learning motivation. The study was conducted at a public university in Turkey with 84 third-year undergraduate nursing students during the 2022-2023 academic year.

Participants were randomly assigned to either the intervention group (n = 42) or the control group (n = 42) using a computer-generated randomization list. The intervention group received the flipped classroom approach, which included:

Access to a specially designed online learning platform with educational videos and reading materials uploaded one week prior to the face-to-face sessions,

A face-to-face session focusing on discussion, case-based learning, and peer interaction led by the researcher,

Learning materials developed based on the "Pediatric Pain Management" content defined in the national nursing education curriculum and international guidelines.

The control group engaged in self-directed learning by studying the same written materials independently without structured guidance or interaction.

Data were collected at three time points:

Pre-test (baseline) before the intervention,

Post-test immediately after the intervention (1 month later),

Follow-up (retention test) three months after the intervention.

Two validated instruments were used:

Pediatric Nurses' Knowledge and Attitudes Survey Regarding Pain (PNKAS) adapted for nursing students to measure knowledge,

Motivation to Learn Scale to assess students' learning motivation.

A two-way mixed ANOVA was used to analyze the effects of the intervention across time and between groups. At baseline, no significant differences were found between groups in either knowledge or motivation scores. However, after the intervention, the intervention group showed statistically significant and sustained improvements in both variables, whereas the control group did not exhibit notable changes.

The findings support the use of the flipped classroom approach as an effective and sustainable educational strategy in nursing education, particularly in areas requiring complex knowledge and critical thinking such as pediatric pain management. Integration of this model into nursing curricula may enhance both cognitive outcomes and motivation to learn.

ELIGIBILITY:
Inclusion Criteria

Being enrolled in the "Child Health and Diseases Nursing" course for the first time

Having access to the Internet and a computer or smartphone

Agreeing to attend synchronous sessions via Google Classroom

Volunteering to participate in the study

Exclusion Criteria

Having previously received any education on pediatric pain management

Withdrawing consent at any point during the study

Failing to complete the pre-test, post-test, or three-month follow-up assessment (e.g., missing a measurement session due to internet connectivity issues)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Pediatric Pain Management Knowledge Score | Baseline (pre-test), 1 month after intervention (post-test), and 3 months after intervention (follow-up)
  The Pediatric Pain Management Knowledge Scale, developed by Aydın & Bektaş (2021), measures nursing students' knowledge of pediatric pain. It consists of 29 items rated on a 5-point Likert scale, covering six sub-dimensions: pain awareness (6 items), pain physiopathology (4), barriers to pain management (11), pain diagnosis (2), pain assessment (2), and pain control (4). Items 3, 6, 8, 10-15, 17, and 21 are reverse coded. Scores range from 29 to 145; higher scores indicate greater knowledge. In this study, Cronbach's alpha was 0.845.

SECONDARY OUTCOMES:
Motivation Level Toward Instructional Materials | Baseline (pre-test), 1 month after intervention (post-test), and 3 months after intervention (follow-up)
  The Motivation Questionnaire for Instructional Materials (MMIM), developed by Keller (2006) and adapted into Turkish by Kutu & Sözbilir (2011), measures students' motivation toward instructional materials. It has 24 items rated on a 5-point Likert scale, with two dimensions: attention-relevance (items 1-11) and confidence-satisfaction (items 12-24). Items 3, 12, 14, 16, and 18 are reverse coded. Scores range from 24 to 120; higher scores indicate higher motivation. Cronbach's alpha was 0.83 in the original study and 0.789 in this study.

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Akif Ersoy University, Faculty of Health Sciences, Burdur, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because participants did not provide consent for external data sharing and the study materials are governed by institutional privacy regulations. Data will remain accessible only to the study team

REFERENCES:
- [Result] Ekim A, Ocakci AF. Knowledge and attitudes regarding pain management of pediatric nurses in Turkey. Pain Manag Nurs. 2013 Dec;14(4):e262-e267. doi: 10.1016/j.pmn.2012.02.004. Epub 2012 Apr 4. PMID 24315279
- [Result] Martin F, Sun T, Westine CD. A systematic review of research on online teaching and learning from 2009 to 2018. Comput Educ. 2020 Dec;159:104009. doi: 10.1016/j.compedu.2020.104009. Epub 2020 Sep 9. PMID 32921895
- [Result] Paralikar S, Shah CJ, Joshi A, Kathrotia R. Acquisition of Higher-Order Cognitive Skills (HOCS) Using the Flipped Classroom Model: A Quasi-Experimental Study. Cureus. 2022 Apr 18;14(4):e24249. doi: 10.7759/cureus.24249. eCollection 2022 Apr. PMID 35602838
- [Result] Zhang D, Huang A, Lei Y, Liu H, Yang L, Wang C, Yuan T, Li X, Zhang L, Shang W. Nursing students' experiences and perceptions regarding in-class flipped classroom: a mixed-methods study. BMC Med Educ. 2025 May 8;25(1):675. doi: 10.1186/s12909-025-07248-x. PMID 40340719
- [Result] Yuan L. Effect of Educational Interventions for Improving the Nurses' Knowledge, Attitude, and Practice of Pediatric Pain Management: A Aystematic Review and Meta-Analysis. Pain Manag Nurs. 2024 Aug;25(4):e271-e278. doi: 10.1016/j.pmn.2024.04.005. Epub 2024 May 3. PMID 38702258
- [Result] Xu P, Chen Y, Nie W, Wang Y, Song T, Li H, Li J, Yi J, Zhao L. The effectiveness of a flipped classroom on the development of Chinese nursing students' skill competence: A systematic review and meta-analysis. Nurse Educ Today. 2019 Sep;80:67-77. doi: 10.1016/j.nedt.2019.06.005. Epub 2019 Jun 14. PMID 31279251
- [Result] Guidelines on the management of chronic pain in children. Geneva: World Health Organization; 2020. Available from http://www.ncbi.nlm.nih.gov/books/NBK566553/ PMID 33433967
- [Result] Ulgen H, Tufekci FG. The Effect of Pain Management Education on Nurses' Pain Knowledge and Attitudes. Pain Manag Nurs. 2024 Jun;25(3):e186-e191. doi: 10.1016/j.pmn.2023.12.011. Epub 2024 Feb 10. PMID 38342705
- [Result] Ung A, Salamonson Y, Hu W, Gallego G. Assessing knowledge, perceptions and attitudes to pain management among medical and nursing students: a review of the literature. Br J Pain. 2016 Feb;10(1):8-21. doi: 10.1177/2049463715583142. Epub 2015 May 13. PMID 27551407
- [Result] Shi, X.-Y., Yin, Q., Wang, Q.-W., Lu, B.-R., Li, G.-X., Huang, S.-H., & Sun, Z.-G. (2025). Is the flipped classroom more effective than the traditional classroom in clinical medical education: A systematic review and meta-analysis. Frontiers in Education, 9, Article 1485540. https://doi.org/10.3389/feduc.2024.1485540
- [Result] Shanmugam SR, Alabdullah AAS, Alenezi MH, Aldughyshim SK, Alnemer MF, Almutairi WK, Alhadyan GS, Albugomi RZ, Alkhulayfi FA. Knowledge and attitudes toward pediatric pain management among nursing interns from a selected university in Riyadh, Saudi Arabia: a descriptive cross-sectional quantitative study. PeerJ. 2025 Apr 21;13:e19288. doi: 10.7717/peerj.19288. eCollection 2025. PMID 40276299
- [Result] Atefeh S. Barriers and facilitators of pain management in children: a scoping review. BMC Anesthesiol. 2025 Apr 1;25(1):148. doi: 10.1186/s12871-025-02941-2. PMID 40170135
- [Result] Shah P, Siu A. Considerations for neonatal and pediatric pain management. Am J Health Syst Pharm. 2019 Sep 16;76(19):1511-1520. doi: 10.1093/ajhp/zxz166. PMID 31504147
- [Result] Raja SN, Carr DB, Cohen M, Finnerup NB, Flor H, Gibson S, Keefe FJ, Mogil JS, Ringkamp M, Sluka KA, Song XJ, Stevens B, Sullivan MD, Tutelman PR, Ushida T, Vader K. The revised International Association for the Study of Pain definition of pain: concepts, challenges, and compromises. Pain. 2020 Sep 1;161(9):1976-1982. doi: 10.1097/j.pain.0000000000001939. PMID 32694387
- [Result] Merrou S, Baslam A, Idrissi Jouicha A, Ouhaz Z, El Adib AR. Blended learning and simulation in nursing education: A quasi-experimental study on a nursing institute. J Educ Health Promot. 2023 Sep 29;12:303. doi: 10.4103/jehp.jehp_72_23. eCollection 2023. PMID 38023106
- [Result] Liu, Y., Li, Y., Lei, M., Liu, P., Theobald, J., Meng, L., Liu, T., Zhang, C., & Jin, C. (2018). Effectiveness of the flipped classroom on the development of self-directed learning in nursing education: A meta-analysis. Frontiers of Nursing, 5, 317-329. https://doi.org/10.1515/fon-2018-0032
- [Result] Liu YM, Lin GL, Chao KY, Jih HJ, Yang BH, Chiang YC. Comparison of the effectiveness of teaching strategies for a pediatric pain management program for undergraduate nursing students: A quantitative evaluation using an objective structured clinical examination. Nurse Educ Pract. 2020 Feb;43:102707. doi: 10.1016/j.nepr.2020.102707. Epub 2020 Jan 18. PMID 31981972
- [Result] Kutu, H., & Sözbilir, M. (2011). Öğretim Materyalleri Motivasyon Anketinin Türkçeye Uyarlanması: Güvenirlik ve Geçerlik Çalışması. Necatibey Faculty of Education Electronic Journal of Science and Mathematics Education, 5(1), 292-312.
- [Result] Keller, J. M. (2006). Development of two measures of learner motivation. In Academy of Human Resource Development International Conference Proceedings (pp. 1063-1070).
- [Result] International Association for the Study of Pain. (2018). IASP curriculum outline on pain for nursing. https://www.iasp-pain.org/education/curricula/iasp-curriculum-outline-on-pain-for-nursing/
- [Result] Gadallah, M. A., Hassan, A. M., Shargawy, S. A. (2017). Undergraduate nursing students' knowledge and attitude regarding pain management of children in Upper Egypt. J Nurs Educ Pract, 7(6), 100-7. https://doi.org/10.5430/jnep.v7n6p100
- [Result] ChildKind International. (2020). Homepage. https://childkindinternational.org/
- [Result] Chen, Y., Wang, Y., Kinshuk, & Chen, N. S. (2014). Is FLIP enough? Or should we use the FLIPPED model instead? Computers & Education, 79, 16-27. https://doi.org/10.1016/j.compedu.2014.07.004
- [Result] Busebaia TJA, Thompson J, Fairbrother H, Ali P. The role of family in supporting adherence to diabetes self-care management practices: An umbrella review. J Adv Nurs. 2023 Oct;79(10):3652-3677. doi: 10.1111/jan.15689. Epub 2023 May 7. PMID 37150951
- [Result] Bond M. Pain education issues in developing countries and responses to them by the International Association for the Study of Pain. Pain Res Manag. 2011 Nov-Dec;16(6):404-6. doi: 10.1155/2011/654746. PMID 22184547
- [Result] Betihavas V, Bridgman H, Kornhaber R, Cross M. The evidence for 'flipping out': A systematic review of the flipped classroom in nursing education. Nurse Educ Today. 2016 Mar;38:15-21. doi: 10.1016/j.nedt.2015.12.010. Epub 2015 Dec 22. PMID 26804940
- [Result] Aydin B, Bektas M. Pediatric Pain Management Knowledge Levels of Intern Nursing Students. Pain Manag Nurs. 2020 Jun;21(3):290-298. doi: 10.1016/j.pmn.2019.06.012. Epub 2019 Aug 8. PMID 31402123
- [Result] WHO Guidelines on the Pharmacological Treatment of Persisting Pain in Children with Medical Illnesses. Geneva: World Health Organization; 2012. Available from http://www.ncbi.nlm.nih.gov/books/NBK138354/ PMID 23720867
- [Result] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Result] 12. Cohen, J. (2013). Statistical power analysis for the behavioral sciences. Routledge. https://doi.org/10.4324/9780203771587
- [Result] Barranquero-Herbosa M, Abajas-Bustillo R, Ortego-Mate C. Effectiveness of flipped classroom in nursing education: A systematic review of systematic and integrative reviews. Int J Nurs Stud. 2022 Nov;135:104327. doi: 10.1016/j.ijnurstu.2022.104327. Epub 2022 Jul 21. PMID 35944288
- [Result] Alshehri FA, Levett-Jones T, Pich J. Nursing students' knowledge of and attitudes towards pain management: An integrative review. Nurse Educ Today. 2024 Aug;139:106207. doi: 10.1016/j.nedt.2024.106207. Epub 2024 Apr 10. PMID 38669861
- [Result] 1. Akdeniz Kudubeş, A., Bektaş, İ., & Bektaş, M. (2021). Nursing role in children pain management. Journal of Education and Research in Nursing, 18(1), 107-113. https://doi.org/10.5152/jern.2021.91489

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-31): https://cdn.clinicaltrials.gov/large-docs/44/NCT07129044/Prot_SAP_000.pdf